CLINICAL TRIAL: NCT07130799
Title: Evaluation of the Innate Immune Response Through Monocyte HLA-DR Monitoring During Severe Intra-abdominal Candidiasis in the Critically Ill Patients
Brief Title: Innate Immune Response Monitoring Via Monocyte HLA-DR in Severe Intra-abdominal Infections at Risk of Fungal Infection
Acronym: CANDIRIS
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024PI208
Record Dates: First submitted 2025-07-24; First posted 2025-08-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Intra-abdominal Infection; Critical Illness; Post-Op Infection; Immunization; Sepsis; Candida Sepsis
Keywords: intra-abdominal infection; intra-abdominal candidiasis; HLA-DR; immunomonitoring; monocyte; critically ill patients
MeSH Terms: conditions — Intraabdominal Infections; Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-abdominal candidiasis: Intra-abdominal infection with intra-abdominal candidiasis based on the FUNDICU consensus
  Interventions: Other: Immunomonitoring
- Bacterial Intra-abdominal infection: Intra-abdominal infection with a negative fungal culture
  Interventions: Other: Immunomonitoring

INTERVENTIONS:
Other: Immunomonitoring — To analyse monocyte HLA-DR expression (mHLA-DR) and CD4+ T lymphocyte count (CD4) in both group

SUMMARY:
Intra-abdominal candidiasis (IAC) is a frequent and severe fungal infection in critically ill patients, often diagnosed late. Its pathophysiology remains unclear, particularly regarding why some patients develop invasive infection while others only show benign colonization. A potential explanation lies in the state of innate immunity. Monocyte HLA-DR expression, a recognized marker of immune suppression in critical care, may be transiently but profoundly reduced in non-immunocompromised patients who go on to develop IAC. This observational study aims to evaluate whether patients with IAC have greater innate immune dysfunction-assessed by HLA-DR expression-compared to those with severe bacterial intra-abdominal infections. The goal is to better understand the immune mechanisms involved and improve early risk stratification for IAC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Patient admitted to the ICU or intermediate care unit for a severe intra-abdominal infection requiring urgent abdominal surgery
* Presence of at least one risk factor for intra-abdominal candidiasis:

  * Abdominal surgery within the last 7 days
  * Supramesocolic gastrointestinal perforation
  * Healthcare-associated intra-abdominal infection
  * Community-acquired intra-abdominal infection in an immunocompromised patient*
  * Intra-abdominal infection complicated by septic shock
  * Broad-spectrum antibiotic exposure within 72 hours prior to surgery
* And/or a Peritonitis Score ≥ 3 out of 4
* Patient affiliated with or benefiting from a national health insurance system
* Patient who has received full information about the clinical study

Exclusion Criteria:

* Radiologically guided drainage without surgery
* Infected acute pancreatitis
* Limitation or withdrawal of life-sustaining treatments
* Moribund patient with an expected life expectancy < 48 hours
* Woman of childbearing potential without effective contraception
* Refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients (≥18 years) admitted to the intensive care unit (ICU) for severe intra-abdominal infections requiring urgent abdominal surgery. Participants must present at least one recognized risk factor for intra-abdominal candidiasis, such as recent abdominal surgery, gastrointestinal perforation, healthcare-associated infection, immunosuppression, septic shock, or recent exposure to broad-spectrum antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between percentage of Monocyte HLA-DR Expression and the Occurrence of Intra-abdominal Candidiasis | Within 7 days after abdominal surgery
  Assessment of the relationship between monocyte HLA-DR expression levels and the development of intra-abdominal candidiasis in critically ill patients with severe intra-abdominal infection.

SECONDARY OUTCOMES:
Change Over Time in Percentage of Monocytes Expressing HLA-DR Measured by Flow Cytometry in Patients With vs Without Intra-abdominal Candidiasis | From Day 0 (surgery) to Day 7 post-surgery
  Peripheral venous blood will be collected at Day 0 (within 6 hours after index surgery), Day 3, Day 5, and Day 7 post-surgery.
  Monocyte HLA-DR expression will be quantified as the percentage of CD14+/CD16-/low monocytes positive for HLA-DR using standardized flow cytometry with anti-HLA-DR monoclonal antibody.
  Results will be compared between patients with confirmed intra-abdominal candidiasis (peritoneal culture positive for Candida) and those with intra-abdominal infection without fungal involvement.
  Primary analysis: between-group difference in change from baseline (Day 0) to Day 7 in percentage of HLA-DR+ monocytes
Variation in Lymphocyte Subpopulations Based on Presence or Absence of Intra-abdominal Candidiasis | From Day 0 (surgery) to Day 7 post-surgery
  Analysis of the changes in lymphocyte subpopulations counts (CD4+ T cells, CD8+ T cells, NK cells, B cells) in patients with versus without intra-abdominal candidiasis
Impact of Immune Dysfunction on In-Hospital Mortality | From surgery to Day 28
  Evaluation of the correlation between low HLA-DR expression and in-hospital mortality
Impact of Immune Dysfunction on Source Control of Infection | Up to 28 days
  Assessment of whether immune dysfunction (defined by a low expression level of HLA-DR) is associated with failure or delay in achieving effective surgical or medical source control of the intra-abdominal infection

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided